CLINICAL TRIAL: NCT07092683
Title: Mediating Role of Intraoperative Red Blood Cell Transfusion in the Relationship Between Preoperative Anaemia and Postoperative Complications in Cardiac Surgery
Brief Title: Mediation Analysis in Cardiac Surgery
Acronym: MACS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20210655
Record Dates: First submitted 2025-07-20; First posted 2025-07-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-07

CONDITIONS: Anemia; Cardiac Surgery; Transfusion; Mediation
MeSH Terms: conditions — Anemia; Negotiating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- anemia
  Interventions: Other: anemia
- nonanemia
  Interventions: Other: nonanemia

INTERVENTIONS:
Other: anemia — preoperative anemia
  Groups: anemia
Other: nonanemia — preoperative nonanemia
  Groups: nonanemia

SUMMARY:
This study investigates the mediating role of intraoperative allogeneic red blood cell transfusion in the relationship between preoperative anaemia and postoperative complications in patients undergoing cardiac surgery. Using mediation analysis methods, we aim to determine whether and to what extent intraoperative transfusion explains the association between preoperative anaemia and adverse postoperative outcomes. By elucidating this pathway, the study seeks to inform perioperative blood management strategies and support more personalized, risk-adapted approaches to minimize postoperative complications in anaemic patients undergoing cardiac procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older ；
* Undergoing elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* preoperative mechanical circulatory support
* ASA physical status VI-V
* unplanned intra-hospital reoperations
* catheter-based valve replacements,
* heart tumours,
* stent implantation surgeries,
* coronary angiography,
* transvascular valve clamping,
* tetralogy of Fallot,
* ventricular aneurysms,
* cardiomyopathies,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients for inclusion were those aged 18 or older undergoing elective cardiac surgery with CPB support at West China Hospital (WCH) from 22 December 2010 to 1 July 2017, and at The Second affiliated Hospital of Zhejiang University (SAHZU) from 1 September 2013 to 31 December 2024.
Sampling Method: Probability Sample
Enrollment: 13683 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications | From the start of surgery to 30 days after surgery
  The primary outcome is the occurrence of any postoperative complications during the index hospitalization. Complications include, but are not limited to, acute kidney injury (AKI), neurological complications, infections, and pulmonary complications. These are assessed using standardized diagnostic criteria.

SECONDARY OUTCOMES:
Incidence of Acute Kidney Injury (AKI) | From the start of surgery to 30 days after surgery
  Occurrence of AKI during postoperative hospitalization, defined according to the KDIGO (Kidney Disease: Improving Global Outcomes) criteria.
Incidence of Neurological Complications | From the start of surgery to 30 days after surgery
  Occurrence of neurological complications such as postoperative delirium, stroke, or cognitive dysfunction, assessed based on clinical diagnosis and relevant neurocognitive evaluation.
Incidence of Infections | From the start of surgery to 30 days after surgery
  Occurrence of postoperative infections including surgical site infection, bloodstream infection, and pneumonia, diagnosed according to CDC criteria.
Incidence of Pulmonary Complications | From the start of surgery to 30 days after surgery
  Occurrence of pulmonary complications including pneumonia, pleural effusion, atelectasis, or need for prolonged mechanical ventilation (>48 hours postoperatively).
Length of Hospital Stay | From the start of surgery to 30 days after surgery
  Duration of postoperative hospital stay, defined as the number of days from the date of surgery to the date of hospital discharge.
Total Hospitalization Cost | From the start of surgery to 30 days after surgery
  Total direct medical cost incurred during the index hospitalization, including surgical costs, intensive care, ward care, medications, laboratory and imaging studies, and blood transfusion-related expenses.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fowler AJ, Ahmad T, Phull MK, Allard S, Gillies MA, Pearse RM. Meta-analysis of the association between preoperative anaemia and mortality after surgery. Br J Surg. 2015 Oct;102(11):1314-24. doi: 10.1002/bjs.9861. PMID 26349842
- [Result] Horvath KA, Acker MA, Chang H, Bagiella E, Smith PK, Iribarne A, Kron IL, Lackner P, Argenziano M, Ascheim DD, Gelijns AC, Michler RE, Van Patten D, Puskas JD, O'Sullivan K, Kliniewski D, Jeffries NO, O'Gara PT, Moskowitz AJ, Blackstone EH. Blood transfusion and infection after cardiac surgery. Ann Thorac Surg. 2013 Jun;95(6):2194-201. doi: 10.1016/j.athoracsur.2012.11.078. Epub 2013 May 3. PMID 23647857
- [Result] Transfusion of Red Blood Cells, Fresh Frozen Plasma, or Platelets Is Associated With Mortality and Infection After Cardiac Surgery in a Dose-Dependent Manner. Anesth Analg. 2020 Feb;130(2):e32. doi: 10.1213/ANE.0000000000004528. PMID 31702696